CLINICAL TRIAL: NCT06234293
Title: Near-Infrared Light Devices Versus Landmark Approach for Peripheral Venous Access in Intensive Care Unit: A Randomized Controlled Study
Brief Title: Near-Infrared Light Devices Versus Landmark Approach for Peripheral Venous Access in Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHRO-2022-14
Record Dates: First submitted 2024-01-15; First posted 2024-01-31 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Upper Limb Edema; Critical Illness
Keywords: Intensive Care Unit; Peripheral Venous Access; Landmark approach; Near-infrared light device; PIVC
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Intervention Model Description: Randomized controlled multicenter trial Ratio 1:1
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- near-infrared light device (Experimental): the device used is the AccuVein AV500® (Accuvein, New York USA). Nurses will have to find the vein for the PIVC using the near-infrared light device. Nurses will have to proceed as follows: apply the tourniquet, put on the near infrared light onto the upper limb. PIVC on the lower limbs is forbidden in this study. The recommended projection distance is around 20 cm, however, the optimal distance of projection can vary between 10 and 45 cm. After finding the vein, Nurses proceed to PIVC with the device turned on, the peripheral venous network visible on the skin of the patient. After the cannulation and to confirm the functionality of the peripheral intravenous access a flash of 10cc of an isotonic solution (NaCl 0.9%) will be injected
  Interventions: Device: near-infrared light device
- landmark approach (No Intervention): PIVC will be done by a nurse on an upper limb according to the standard approach. The nurse will proceed as follows: apply the tourniquet and find a vein for the catheterization, standard techniques to highlight veins can be used (apply alcohol, tap veins …). After finding a vein, the nurses proceed to the PIVC according to his / her habits. The use of any device is forbidden. After the cannulation and to confirm the functionality of the peripheral venous access a flash of 10cc of an isotonic solution (NaCl 0.9%) will be injected.

INTERVENTIONS:
Device: near-infrared light device — Nurses will have to find the vein for the PIVC using the near-infrared light device.
  Arms: near-infrared light device

SUMMARY:
The central venous catheter (CVC) is commonly used in intensive care unit (ICU). The primary complications associated with CVCs especially with prolonged use include thrombosis and infections. Hence, it is essential to remove the CVC as soon as it becomes unnecessary.

Peripheral intravenous cannulation (PIVC) on a critically ill patient can be a significant challenge for nurses. After several days in ICU, patients may develop significant edema in the upper limbs, complicating the PIVC.

Near-infrared light devices (NILD) are medical devices that use near-infrared light to highlight the patient's peripheral venous network directly on their skin. The advantage of this device is its minimal training and ease of use for effective application. Nurses can use this medical device without specific conditions once they have received training on its use. The vein illuminator has not been extensively studied in ICU.

This study aims to compare two techniques for PIVC in critically ill patients with existing CVC for whom maintaining the deep venous access is no longer indicated.

The investigators hypothesize that the use of the NILD would increase the success rate of first-attempt PIVC insertion compared to a landmark approach (traditional method) for PIVC in ICU.

DETAILED DESCRIPTION:
This is a multicenter randomized controlled study. 380 patients will be randomly assigned with a 1:1 ratio to landmark approach (standard group) or near-infrared light device (interventional group).

Randomization will be done immediately after the enrollment of the patient. Randomization will be stratified by center and according to anticipated difficult venous access defined by:

* BMI > 30 Kg/m2
* Increase in body weight between admission and day of inclusion > 10%.
* Clinically evident edema of the upper limbs (with pitting)
* Absence of visible or palpable veins on arms and forearms If one or more items are present, the patient is classified as difficult to venous access.

Once the patient has been enrolled and randomized, the nurse in charge of the patient performs the PIVC according to the randomization group as soon as possible after randomization.

The nurse will have a maximum of 3 attempts before handing over to another nurse. The total number of attempts will be 5 with the allocated method (traditional method or NILD).

In the case of failure after 5 initial attempts, the intervention will be considered as a failure. However, a maximum of 5 additional attempts will be allowed with any method on the day of randomization. The success or failure of PIVC will be recorded, as well as the device used. The attempts should be performed within 6 hours after randomization.

If one of the 5 first initial attempts is successful, the study continues until the PIVC is removed (max 7 days according to recommendations) or patient discharge, whichever comes first, in order to evaluate the occurrence of local complications.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Hospitalized in ICU
* with a deep venous catheter (jugular, subclavian or femoral)
* In whom the use of a deep venous line is no longer justified (absence of: vasopressor amines, chemotherapy, parenteral nutrition, hypertonic solutions)

Exclusion Criteria:

* Absolute contraindication or anatomical impossibility to perform a PIVC on the upper limbs
* Patient already included in the study
* Tattoo covering most of both forearms
* Adult subject to a legal protection measure (guardianship, curators, person under court protection)
* Persons deprived of their liberty by a judicial or administrative decision, persons hospitalised without consent and persons admitted to a health or social establishment for purposes other than research.
* Pregnant or breast-feeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2024-02-28 (Actual); Primary Completion 2025-07-09 (Actual); Study Completion 2025-07-16 (Actual)

PRIMARY OUTCOMES:
Success rate on the first attempt of PIVC in ICU using NILD | Baseline
  To show that the use of the NILD improves the success rate on the first attempt of PIVC in ICU for patients for whom the use of a deep venous catheter is no longer justified.
  The success of PIVC will be determined by the presence of venous return during catheterization in the reflux chamber, the full catheter introduction, and the administration of a 10cc syringe of isotonic solution (NaCl 0.9%) with a flash without extravasation. A puncture attempt is defined by the effraction of the skin barrier by the device.
  During a puncture, repositioning/change of catheter direction is permitted. Peripheral intravenous puncture will be performed by nurses only.

SECONDARY OUTCOMES:
number of attempts before successful PIVC | Baseline
  Compare the number of attempts before successful PIVC between the traditional method (standard group) and the use of NILD (interventional group).
  The number of puncture attempts will be defined by the number of attempts between inclusion and successful of PIVC (last attempt included). On the day of inclusion in the study, each nurse has a maximum of three attempts at PIVC, per patient, depending on the randomization arm. The maximum number of initial attempts per patient is 5.
occurrence of local complications | Day 7
  Compare the occurrence of local complications (phlebitis, extravasation) between the two groups in patients for whom PIVC is considered successful.
  - The occurrence and type of local complications within 7 days of successful PIVC will be compared between the two groups, as well as their time of occurrence after placement (until removal of the medical device or until discharge from the hospital department). if the patient is discharged before 7 days).
  The main local complications are venous inflammation and extravasation. Local signs to watch out for include pain, swelling and induration. The presence of any of these signs during daily monitoring will lead to its withdrawal. Only medical confirmation of venous inflammation and extravasation will be recorded for this study.
success rate of PIVC according to nurses's experience | Baseline
  Compare the success rate of PIVC according to nurses' experience between the two groups.
  The success rate or PIVC according to nurses-experience between the two groups will be compared by stratification: nurses with less than one year's nursing experience, between 1 to 5 years' experience and more than 5 years.
success rate of PIVC in patients considered with anticipated difficult intravenous access | Baseline
  Compare the success rate of PIVC in patients considered with anticipated difficult intravenous access between the two groups.
  - Anticipated difficult PIVC will be defined as follows:
  * Presence of upper limb edema
  * Absence of palpable veins when applying a tourniquet
  * Obese patient defined as BMI > 30 kg/m2
  * Increase in body weight between admission and day of inclusion > 10%
PIVC insertion time | Baseline
  Compare PIVC insertion time between the two groups
pain levels | Baseline
  Compare pain levels in conscious patients between the two groups using the pain verbal analog scale from 0 to 10, where 0 is no pain and 10 unbearable pain.

CONTACTS AND LOCATIONS:
Overall Officials: Aude FERRIER, Principal Investigator — CHU Orléans
Locations (4):
- France (4):
  - CH de Chartres, Chartres
  - CH Le Mans, Le Mans
  - CHU Orléans, Orléans
  - CHU de Tours, Tours

REFERENCES:
- [Background] Gregg SC, Murthi SB, Sisley AC, Stein DM, Scalea TM. Ultrasound-guided peripheral intravenous access in the intensive care unit. J Crit Care. 2010 Sep;25(3):514-9. doi: 10.1016/j.jcrc.2009.09.003. Epub 2009 Oct 15. PMID 19836193
- [Background] Carr PJ, Rippey JCR, Cooke ML, Trevenen ML, Higgins NS, Foale AS, Rickard CM. Factors associated with peripheral intravenous cannulation first-time insertion success in the emergency department. A multicentre prospective cohort analysis of patient, clinician and product characteristics. BMJ Open. 2019 Apr 2;9(4):e022278. doi: 10.1136/bmjopen-2018-022278. PMID 30944127
- [Background] Bridey C, Thilly N, Lefevre T, Maire-Richard A, Morel M, Levy B, Girerd N, Kimmoun A. Ultrasound-guided versus landmark approach for peripheral intravenous access by critical care nurses: a randomised controlled study. BMJ Open. 2018 Jun 9;8(6):e020220. doi: 10.1136/bmjopen-2017-020220. PMID 29886442
- [Background] Curtis SJ, Craig WR, Logue E, Vandermeer B, Hanson A, Klassen T. Ultrasound or near-infrared vascular imaging to guide peripheral intravenous catheterization in children: a pragmatic randomized controlled trial. CMAJ. 2015 May 19;187(8):563-570. doi: 10.1503/cmaj.141012. Epub 2015 Apr 20. PMID 25897047
- [Background] Park JM, Kim MJ, Yim HW, Lee WC, Jeong H, Kim NJ. Utility of near-infrared light devices for pediatric peripheral intravenous cannulation: a systematic review and meta-analysis. Eur J Pediatr. 2016 Dec;175(12):1975-1988. doi: 10.1007/s00431-016-2796-5. Epub 2016 Oct 26. PMID 27785562
- [Derived] Ferrier A, Despres A, Brasselet A, Badre G, Wanneveich M, Nay MA. Near-infrared light devices versus landmark approach for peripheral venous access in the intensive care unit: protocol of a randomised controlled study. BMJ Open. 2025 Aug 18;15(8):e102390. doi: 10.1136/bmjopen-2025-102390. PMID 40829834